CLINICAL TRIAL: NCT03709823
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 2b Trial of Cytisine in Adult Smokers
Brief Title: Trial of Cytisine in Adult Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-CYT-09
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1.5 mg Cytisine, Commercial Schedule (Experimental): 1.5 mg cytisine dose using the commercial 25-day titration schedule + behavioral support
  Interventions: Drug: Cytisine; Behavioral: Behavioral support
- 3.0 mg Cytisine, Commercial Schedule (Experimental): 3.0 mg cytisine dose using the commercial 25-day titration schedule + behavioral support
  Interventions: Drug: Cytisine; Behavioral: Behavioral support
- Placebo, Commercial Schedule (Placebo Comparator): Placebo tablets using the commercial 25-day titration schedule + behavioral support
  Interventions: Drug: Placebo Comparator; Behavioral: Behavioral support
- 1.5 mg Cytisine, TID Schedule (Experimental): 1.5 mg cytisine dose for 25 days using a simplified 3 times daily (TID) schedule + behavioral support
  Interventions: Drug: Cytisine; Behavioral: Behavioral support
- 3.0 mg Cytisine, TID Schedule (Experimental): 3.0 mg cytisine dose for 25 days using a simplified TID schedule + behavioral support
  Interventions: Drug: Cytisine; Behavioral: Behavioral support
- Placebo, TID Schedule (Placebo Comparator): Placebo tablets for 25 days using a simplified TID schedule + behavioral support
  Interventions: Drug: Placebo Comparator; Behavioral: Behavioral support

INTERVENTIONS:
Drug: Cytisine — film coated tablet containing 1.5 mg cytisine in a single tablet
  Arms: 1.5 mg Cytisine, Commercial Schedule; 1.5 mg Cytisine, TID Schedule; 3.0 mg Cytisine, Commercial Schedule; 3.0 mg Cytisine, TID Schedule
Drug: Placebo Comparator — 1.5 mg cellulose powder to match final weight of the cytisine tablet
  Arms: Placebo, Commercial Schedule; Placebo, TID Schedule
Behavioral: Behavioral support — 12 behavioral support sessions by a qualified staff member plus supportive literature and online resources

SUMMARY:
This placebo-controlled Phase 2b trial is being conducted at sites within the United States (US) to evaluate the effectiveness cytisine dosage (1.5 mg, 3.0 mg) and administration schedule (commercial titration versus simplified 3 times daily [TID] schedule) within a 25-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age ≥ 18 years.
2. Current daily cigarette smokers (averaging ≥ 10 cigarettes per day upon completing a 7-day screening diary) and who intend to quit smoking.
3. Expired air carbon monoxide (CO) ≥ 10 parts per million (ppm).
4. Failed at least one previous attempt to stop smoking with or without therapeutic support.
5. Willing to initiate study treatment on the day after randomization and set a quit date that is 5-7 days after starting treatment.
6. Willing to actively participate in the study's smoking cessation behavioral support provided throughout the study.
7. Able to fully understand all study requirements, willing to participate, comply with dosing schedule, and sign the Informed Consent Form.

Exclusion Criteria:

1. Known hypersensitivity to cytisine or any of the excipients.
2. Positive urinary drugs of abuse screen, determined within 28 days before the first dose of cytisine.
3. Clinically significant abnormal serum chemistry or hematology values within 28 days of randomization (i.e. requiring treatment).
4. Clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined after minimum of 5 minutes in supine position within 28 days of randomization (i.e. requiring treatment or further assessment).
5. Body mass index (BMI) classification for being underweight (< 18.5 kg/m^2) or having ≥ Class 2 obesity (≥ 35 kg/m^2).
6. Recent history (within 3 months) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident or hospitalization for congestive heart failure.
7. Current uncontrolled hypertension (blood pressure ≥ 160/100 mmHg).
8. Documented diagnosis of schizophrenia or bipolar psychiatric illness; currently psychotic; having suicidal ideation (Suicide Behaviors Questionnaire-Revised [SBQ-R] score ≥ 7); or current symptoms of moderate to severe depression (Hospital Anxiety and Depression Scale [HADS] score ≥ 11).
9. Renal impairment defined as a creatinine clearance (CrCl) < 60 mL/min (estimated with the Cockroft-Gault equation) or hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.0 times the upper limit of normal (ULN).
10. Women who are pregnant or breast-feeding.
11. Male or Female subjects of child bearing potential who do not agree to use acceptable methods of birth control during the study treatment period.
12. Participation in a clinical study with an investigational drug within 4 weeks of randomization.
13. Treatment with other smoking cessation medications (bupropion, varenicline, nortriptyline, or any nicotine replacement therapy [NRT]) within 4 weeks of randomization or planned use of these other smoking cessation medications during the study.
14. Use within 2 weeks of randomization or planned use during the study of non-cigarette nicotine products (e-cigarettes, pipe tobacco, cigars, snuff, chewing tobacco, hookah) or marijuana vaping or smoking.
15. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Nides, PhD, Principal Investigator — Los Angeles Clinical Trials
Locations (8):
- United States (8):
  - Clinical Research Consortium, Tempe, Arizona
  - Los Angeles Clinical Trials, Burbank, California
  - Central Kentucky Research Associates, LLC, Lexington, Kentucky
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Rochester Clinical Research, Inc, Rochester, New York
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - FutureSearch Trails of Dallas, LP, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1.5 mg Cytisine, Commercial Schedule | 3.0 mg Cytisine, Commercial Schedule | Placebo, Commercial Schedule | 1.5 mg Cytisine, TID Schedule | 3.0 mg Cytisine, TID Schedule | Placebo, TID Schedule
Started | 51 | 50 | 25 | 52 | 50 | 26
Completed | 48 | 45 | 22 | 50 | 49 | 26
Not Completed | 3 | 5 | 3 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Other, Not Specified | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1.5 mg Cytisine, TID Schedule: 1.5 mg cytisine dose for 25 days using a simplified TID schedule + behavioral support
- Total: Total of all reporting groups
Arm/Group | 1.5 mg Cytisine, Commercial Schedule | 3.0 mg Cytisine, Commercial Schedule | Placebo, Commercial Schedule | 1.5 mg Cytisine, TID Schedule | 3.0 mg Cytisine, TID Schedule | Placebo, TID Schedule | Total
Number analyzed (Participants) | 51 | 50 | 25 | 52 | 50 | 26 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.46) | 50.0 (13.20) | 51.0 (15.16) | 47.0 (13.67) | 46.3 (12.88) | 47.0 (12.64) | 48.4 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 14 | 29 | 25 | 17 | 133
  Male | 23 | 30 | 11 | 23 | 25 | 9 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 3 | 13 | 7 | 7 | 46
  White | 43 | 40 | 21 | 37 | 41 | 18 | 200
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 2 | 6 | 1 | 0 | 15
  Not Hispanic or Latino | 45 | 49 | 23 | 46 | 49 | 26 | 238
  Native American | 1 | 0 | 0 | 0 | 0 | 0 | 1
Average Number of Cigarettes Smoked per Day Over 7 Consecutive Days [Mean (Standard Deviation); unit: cigarettes per day] — As reported in the participant's 7-day diary, which was completed between screening visits 1 and 2.
  cigarettes per day | 17.6 (5.30) | 18.0 (5.51) | 16.7 (4.28) | 18.0 (6.69) | 18.0 (6.12) | 18.0 (5.96) | 17.8 (5.75)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Analysis of Primary Outcome Measure: Percentage of Expected Cigarettes Smoked Per Participant During Study Treatment
Description: The daily cigarette counts (number of cigarettes smoked in the past 24 hours) were self-reported by participants in the diary. Percentage of expected cigarettes smoked was computed for each participant at the end of treatment (cigarette score), based on daily cigarette counts during treatment vs the screening period. The percentage of expected cigarettes smoked was computed as Y = (100 x N) / (T x R) where N represents total number of cigarettes smoked each day over the treatment period from Day 1 to Day 25; T represents number of post-randomization days where number of cigarettes smoked is recorded; and R represents the average number of cigarettes smoked daily over the 7-day screening period as baseline. T*R represents the total number of cigarettes that would have been smoked without intervention over the number of recorded days. Separate statistical analyses were performed for the two cytisine administration schedules (commercial and TID).
Time Frame: Day 1 through Day 25
Measure: Least Squares Mean (Standard Error); unit: percentage of cigarettes smoked
Arm/Group | 1.5 mg Cytisine, Commercial Schedule | 3.0 mg Cytisine, Commercial Schedule | Placebo, Commercial Schedule | 1.5 mg Cytisine, TID Schedule | 3.0 mg Cytisine, TID Schedule | Placebo, TID Schedule
Number analyzed (Participants) | 51 | 50 | 25 | 52 | 50 | 26
percentage of cigarettes smoked | 26.62 (3.085) | 25.04 (3.123) | 47.10 (4.417) | 29.40 (3.046) | 32.50 (3.105) | 35.30 (4.392)
Statistical Analysis 1: Comparison: 1.5 mg Cytisine, Commercial Schedule vs Placebo, Commercial Schedule; Test type: Superiority; p = 0.0002, ANOVA — Based on analysis of variance models with percent of expected cigarettes smoked as the dependent variable, treatment and body mass index class as main fixed effects, with covariate of baseline cigarettes; LS Mean Difference vs. Placebo = -20.48, 95% CI 2-sided [-31.141 to -9.821]
Statistical Analysis 2: Comparison: 3.0 mg Cytisine, Commercial Schedule vs Placebo, Commercial Schedule; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -22.07, 95% CI 2-sided [-32.791 to -11.342]
Statistical Analysis 3: Comparison: 1.5 mg Cytisine, TID Schedule vs Placebo, TID Schedule; Test type: Superiority; p = 0.2708, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -5.90, 95% CI 2-sided [-16.463 to 4.660]
Statistical Analysis 4: Comparison: 3.0 mg Cytisine, TID Schedule vs Placebo, TID Schedule; Test type: Superiority; p = 0.6018, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -2.81, 95% CI 2-sided [-13.438 to 7.820]
Statistical Analysis 5: Comparison: Placebo, Commercial Schedule vs Placebo, TID Schedule; Test type: Superiority; p = 0.1025, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Commercial Sched. = -12.17, 95% CI 2-sided [-26.869 to 2.535]

2. Primary Outcome: Sensitivity Analysis of Primary Outcome Measure: Analysis for Percentage of Expected Cigarettes Smoked Versus Pooled Placebo Arms, Commercial Schedule
Description: The daily cigarette counts (number of cigarettes smoked in the past 24 hours) were self-reported by participants in the diary. Percentage of expected cigarettes smoked was computed for each participant at the end of treatment (cigarette score), based on daily cigarette counts during treatment vs the screening period. (See Outcome Measure 1 description for details.) The sensitivity analysis of the primary outcome measure was only performed if results of "Statistical Analysis 5" for Outcome Measure 1 demonstrated the placebo treatment arms (commercial and TID) were not significantly different, and so could be pooled. Separate statistical analyses were performed for the two cytisine administration schedules (commercial and TID).
Time Frame: Day 1 through Day 25
Measure: Least Squares Mean (Standard Error); unit: percentage of expected cigarettes smoked
Groups:
- Pooled Placebo: Placebo tablets using the commercial 25-day titration schedule + behavioral support pooled with Placebo tablets for 25 days using a simplified TID schedule + behavioral support
Arm/Group | 1.5 mg Cytisine, Commercial Schedule | 3.0 mg Cytisine, Commercial Schedule | Pooled Placebo
Number analyzed (Participants) | 51 | 50 | 51
percentage of expected cigarettes smoked | 26.68 (3.065) | 25.08 (3.100) | 41.29 (3.099)
Statistical Analysis 1: Comparison: 1.5 mg Cytisine, Commercial Schedule vs Pooled Placebo; Test type: Superiority; p = 0.0010, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -14.61, 95% CI 2-sided [-23.216 to -6.009]
Statistical Analysis 2: Comparison: 3.0 mg Cytisine, Commercial Schedule vs Pooled Placebo; Test type: Superiority; p = 0.0003, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -16.20, 95% CI 2-sided [-24.862 to -7.548]

3. Primary Outcome: Sensitivity Analysis of Primary Outcome Measure: Analysis for Percentage of Expected Cigarettes Smoked Versus Pooled Placebo Arms, TID Schedule
Description: as for outcome 2
Time Frame: Day 1 through Day 25
Measure: Least Squares Mean (Standard Error); unit: percentage of expected cigarettes smoked
Arm/Group | 1.5 mg Cytisine, TID Schedule | 3.0 mg Cytisine, TID Schedule | Pooled Placebo
Number analyzed (Participants) | 52 | 50 | 51
percentage of expected cigarettes smoked | 29.29 (3.291) | 32.41 (3.355) | 41.71 (3.358)
Statistical Analysis 1: Comparison: 1.5 mg Cytisine, TID Schedule vs Pooled Placebo; Test type: Superiority; p = 0.0091, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -12.41, 95% CI 2-sided [-21.695 to -3.135]
Statistical Analysis 2: Comparison: 3.0 mg Cytisine, TID Schedule vs Pooled Placebo; Test type: Superiority; p = 0.0518, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference vs. Placebo = -9.30, 95% CI 2-sided [-18.667 to 0.075]

ADVERSE EVENTS:
Time Frame: From 1st dose of study drug through Week 8 (± 3 days) post-randomization
Arm/Group | 1.5 mg Cytisine, Commercial Schedule | 3.0 mg Cytisine, Commercial Schedule | Placebo, Commercial Schedule | 1.5 mg Cytisine, TID Schedule | 3.0 mg Cytisine, TID Schedule | Placebo, TID Schedule
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/25 | 0/52 | 0/50 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/25 | 0/52 | 0/50 | 0/26
Other Adverse Events (participants affected / at risk) | 16/51 | 16/50 | 5/25 | 15/52 | 14/50 | 8/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg Cytisine, Commercial Schedule (N=51) | 3.0 mg Cytisine, Commercial Schedule (N=50) | Placebo, Commercial Schedule (N=25) | 1.5 mg Cytisine, TID Schedule (N=52) | 3.0 mg Cytisine, TID Schedule (N=50) | Placebo, TID Schedule (N=26)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 1 | 1 | 3 | 4
Fatigue (General disorders) | 1 | 2 | 1 | 3 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3 | 5 | 3 | 4
Headache (Nervous system disorders) | 1 | 1 | 0 | 6 | 2 | 2
Abnormal dreams (Psychiatric disorders) | 4 | 7 | 1 | 4 | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 4 | 1 | 4 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT03709823/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT03709823/SAP_001.pdf